CLINICAL TRIAL: NCT00135200
Title: A Phase II Clinical Trial of Consolidation Treatment With Iodine I 131 Tositumomab for Multiple Myeloma
Brief Title: Clinical Trial of Consolidation Treatment With Iodine I 131 Tositumomab for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2005.035; IRB # 2005-0403 and HUM 43767 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bexxar therapeutic (Experimental): The Bexxar therapeutic regimen is delivered in two sets of intravenous infusions given 7-14 days apart. Nonradioactive Tositumomab is given before both the "dosimetric" infusion and the "therapeutic" infusion to improve distribution of these doses throughout the body. A trace amount of radioactive Iodine 131 Tositumomab is initially given to enable physicians to evaluate the clearance of radiation from the subject's body with gamma camera scans. Calculations made on the basis of these individualized radiation clearance rates allow the therapeutic dose (given 7-14 days after the dosimetric infusion) to be tailored for each patient. The therapeutic dose contains Tositumomab labeled with the amount of Iodine 131 tositumomab specifically calculated based on the scans performed following the dosimetric dose.
  Interventions: Drug: Iodine I 131 Tositumomab

INTERVENTIONS:
Drug: Iodine I 131 Tositumomab — The Bexxar therapeutic regimen is delivered in two sets of intravenous infusions given 7-14 days apart. Nonradioactive Tositumomab is given before both the "dosimetric" infusion and the "therapeutic" infusion to improve distribution of these doses throughout the body. A trace amount of radioactive Iodine 131 attached to Tositumomab is initially given to enable physicians to evaluate the clearance of radiation from your body with gamma camera scans. Calculations made on the basis of these individualized radiation clearance rates allow the therapeutic dose (given 7-14 days after the dosimetric infusion) to be tailored for each patient. The therapeutic dose contains Tositumomab labeled with the amount of Iodine 131 tositumomab specifically calculated for you based on the scans performed following the dosimetric dose.
  Other Names: Bexxar

SUMMARY:
This study is for patients with newly diagnosed or relapsed multiple myeloma. The main purpose of this study is to see how their disease responds to consolidation treatment (treatment aimed at further decreasing cancer cells) with a radioactive antibody (protein) called iodine I 131 tositumomab (known by the tradename Bexxar®) and also to look at the side effects which occur with this type of treatment. The investigators will also be looking at how long disease responds to treatment, if it responds at all, and how long patients who have had this treatment survive.

Bexxar is a monoclonal antibody (protein) to which radioactive iodine 131 is attached. The monoclonal antibody in Bexxar (tositumomab), targets a protein called CD20 found on the surface of a variety of B-cells, including lymphoma cells, and some myeloma cells. The antibody is given as an infusion and finds its way to these cells. The radioactive iodine attached to the antibody delivers radiation directly to these cells which works to harm or kill the cancer cells. Approximately 20-25% of patients with multiple myeloma have this protein on the surface of their tumor cells. In addition, this protein was found on the surface of myeloma stem cells. While myeloma stem cells represent a minority of all myeloma cells (less than 5%), these cells are resistant to chemotherapy and are believed to be responsible for a recurrence of the disease after chemotherapy. In this study, Bexxar will be used after patients complete a course of chemotherapy and have residual myeloma cells left in their body. The Investigators are hoping that the treatment with Bexxar will decrease and possibly eliminate residual myeloma cells resistant to chemotherapy.

DETAILED DESCRIPTION:
Multiple myeloma is ranked second in hematological malignancies in the United States (Munshi et al., 2001). Because no curable option exists, patients with early stage disease are typically observed without treatment until the disease progresses or symptoms appear.

The majority of patients will respond to initial chemotherapy, however, all treated patients repeatedly relapse with shorter remissions following each subsequent course of chemotherapy (Rajkumar et al., 2002a). Regimens most commonly used for initial therapy include melphalan and prednisone (MP), which induce remission in approximately 50% of patients (Alexanian et al., 1969), VAD-vincristine, adriamycin and dexamethasone with response rates in the 50% range (Salmon et al., 1994; Barlogie et al., 1984; Alexanian et al., 1986), dexamethasone pulses, and more recently introduced combinations of thalidomide with dexamethasone (Rajkumar et al., 2002b; Weber et al., 2003). All these regimens have comparable response rates. With the exception of the recent report, which showed a superior response rate to the combination of thalidomide with dexamethasone versus dexamethasone pulses (Rajkumar et al., 2004), multiple other comparative studies did not show superiority of any of these regimens for overall survival. Complete responses to any of these regimens are observed infrequently (< 5%). Patients who complete initial therapy, usually proceed to high dose chemotherapy with autologous stem cell transplant support. Alternatively, patients may be placed on maintenance regimen or can be observed. Except for one study with alternate day high dose of Prednisone (Berenson et al., 2002), no convincing evidence exists that maintenance impacts the natural history of the disease (Kyle, 2002; The Myeloma Trialists' Collaborative Group, 2001).

High dose chemotherapy has been used as consolidation in multiple myeloma by a number of investigators (Barlogie et al., 1986; Cunningham et al., 1994; Harousseau et al., 1995). A randomized trial conducted by French Myeloma Intergroup (IFM 90) provided evidence that treatment with high dose chemotherapy and autologous stem cell transplant (ASCT) after initial therapy results in significantly longer event-free survival (median 28 vs. 18 months) and overall survival (57 vs. 42 months) if compared to conventional chemotherapy (Attal et al., 1996). The benefit of auto transplantation was seen in patients of all ages (Siegel et al., 1999). More recently, similar results were reported from a large randomized study in Great Britain (Childs et al., 2003). Based on these studies, in patients eligible for transplant, consolidation of initial therapy with high dose therapy followed by ASCT is considered a standard of care (NCCN Guidelines 2004). However, ASCT is not curative even in patients who achieve complete response (CR), which is observed in 20-30% of patients who completed ASCT. Contamination of autologous stem cell collection with malignant myeloma cells may play some role. In support of this notion, syngeneic bone marrow transplants showed better and more durable outcomes than those seen with ASCT (Gahrton et al., 1999). Another reason for failure of autologous stem cell transplant is ineffective eradication of myeloma clone with high dose chemotherapy. In an effort to provide more effective elimination of malignant clones, some investigators developed intensified treatment regimens. Improved results have been reported using Total Therapy, which involves a sequence of treatments, including tandem ASCT (Barlogie et al., 1999, Barlogie at al., 2004). The notion that intensification of therapy improves outcomes has been validated in a recent randomized study, which showed that consolidation of initial therapy with tandem autologous stem cell transplant was superior than consolidation with single autologous stem cell transplant as measured by an improved duration of responses and overall survival (Attal at al, 2003). In contrast to ASCT, allogeneic stem cell transplantation can provide stem cell products free of malignant cells, as well as the benefit of graft-versus-myeloma effect.

However, very high 1-year mortality (30-60%) was reported in early allogeneic bone marrow transplant studies, with disease free survival in only 15-30% of patients and no superior survival if compared to ASCT (Bensinger et al., 1996; Bjorkstrand et al., 1996; Barlogie et al., 1995). More recent studies, including allogeneic transplants with nonmyeloablative conditioning regimens, provide more encouraging results (Reynolds et al., 2001; Badros et al., 2002). Recently, a combined treatment with ASCT followed by a non-myeloablative allogeneic stem cell transplant showed very promising outcomes and improved, although still significant toxicity, with CR rates in 55-60% range (Kroger et al., 2002; Maloney et al., 2003). It is too early to determine whether improved responses using this approach will result in an increased survival.

Emerging data suggest that achieving CR or near CR (nCR) will result in more durable remission and longer survival. Recent analysis of long term outcomes of patients treated on randomized French study IMG90 clearly indicates that the longest survivors are those patients who achieve at least very good partial response or complete response (Harousseau, 2003). At 7 years, 60% of patients were alive in a group, which achieved CR or near CR. In contrast, in a group of patients who achieved > PR but less than CR or near CR only 30% were alive and among patients who had less than PR none were alive. Similar results have bee recently reported for patients who underwent allogeneic stem cell transplant (Corradini et al., 2003). It is not clear whether CR in response to initial therapy and prior to transplant may have similar impact on overall outcomes. Regardless of specific transplant approach, survival curves do not plateau and all patients are expected to relapse, regardless of method of intensification therapy, possibly due to persistence of residual population of chemotherapy-resistant clonogenic myeloma cells.

For patients who have relapsed or are refractory to therapy, there is no agreed upon standard treatment (Anderson et al., 2002; Kyle, 2002). Treatment options include salvage chemotherapy, autologous stem cell transplant (if not previously done or as a second transplant), or allogeneic stem cell transplant, full or low intensity (Kyle, 2002). Salvage chemotherapy is most widely used in clinical practice. Among a variety of salvage regimens, both monotherapy and combination therapy have been applied. Monotherapy with Dexamethasone or other steroids administered as pulse therapy produced responses in the 35-40% range (Alexanian et al., 1983; Gertz et al., 1995). Thalidomide used as a single agent showed a 32% response rate in this patient population (Singhal et al., 1999). More recently, VELCADE as a single agent induced at least minimal responses (i.e. > 25% reduction in monoclonal protein) in 35% of patients and at least a stabilization of the disease in 59% of patients with relapsed/refractory multiple myeloma using strict SWOG criteria (Richardson et al., 2003). Combination therapies historically show higher response rates. VAD has been demonstrated as an effective regimen in patients refractory to alkylating agents, with response rates of 60% (Lokhorst et al., 1989). A similar regimen called DVd, with Doxil, Vincristine, and dexamethasone, showed comparable efficacy and acceptable toxicity (Hussein et al., 2002; Rifkin et al., 2004). Newer combinations, including combinations of VELCADE, thalidomide, and Revlimid (analog of thalidomide) are promising, and appear to be able to induce higher response rates and complete remissions as per unpublished yet reports from different meetings (Agarwal et al, 2003; Orlowski et al, 2003, Richardson et al, 2003; Richardson et al., 2004).

Clonogenic Multiple Myeloma Cells:

Myeloma is characterized by an accumulation of malignant plasma cells in bone marrow. Numerous observations indicated that malignant plasma cells have low proliferative capacity and it is believed that the vast majority of the malignant cell population in myeloma is represented by terminally differentiated plasma cells, similar to their normal counterparts (Barlogie et al., 1989). It is unclear whether these terminally differentiated malignant plasma cells are capable of self-renewal. During the past decade, several studies indicated that multiple myeloma, similarly to other malignancies, may consist of heterogenous population of malignant cells (Bakkus et al., 1994; Billadeau et al., 1996).

Clonotypic studies identified a population of circulating B-cells in blood samples of patients with myeloma (Bergsagel et al., 1995, Chen and Epstein, 1996), sharing the same clonotypic CDR3 region as is detected in the bone marrow malignant plasma cells (Pilarski et al, 1996, Szczepek et al., 1998). Further studies provided additional insights into the evolution of the myeloma clone supporting a notion of heterogeneity of the population of clonal cells in myeloma (Taylor et al., 2002). The B-cell component of the myeloma clone appeared to be clonogenic in xenografted mice (Pilarski et al., 2000; Reiman et al., 2001). Moreover, clonotypic cells with B-cell phenotype express CD19+/CD20+ antigens and may represent a reservoir of disease that persists after therapy, including high dose chemotherapy (Kiel et al., 1999; Rottenburger et al., 1999; Pilarski et al., 2002).

The majority of myeloma cells express CD138, a highly specific surface antigen of terminally differentiated plasma cells, which is absent on highly proliferative normal plasmablast and earlier stages of B-cells (Jego et al., 2001). Based on these observations, it was hypothesized that clonogenic myeloma cells should lack CD138 expression. Using CD138+ and CD138- subsets of cells isolated from myeloma cell lines and from primary myeloma patient samples, Matsui et al. (2004), showed that only a minority of all myeloma cells have CD138- phenotype (<5%). However, only CD138- have clonogenic potential, as demonstrated in colony formation assays in methylcellulose and after transplantation to NOD/SCID mice. Moreover, these cells express B-cell antigens, including CD19 and CD20 and their growth could be inhibited by in vitro treatment with rituximab, an antibody directed against CD20 antigen (Matsui et al., 2004).

Rationale for anti-CD20 Therapy in Myeloma:

Recent observations that clonogenic cells in myeloma express CD20 (Kiel et al, 1999, Rottenburger et al, 1999) and that their growth could be inhibited in vitro by rituximab, an anti-CD20 antibody (Matsui et al, 2004), provides a rationale for using CD20-directed therapy in patients with myeloma. Moreover, CD19+/CD20+ clonotypic cells appear to be more refractory than CD19-/CD20- cells to commonly used chemotherapy regimens in myeloma including high dose therapy with stem cell transplant (Kiel et al., 1999, Rottenburger et al, 1999). Therefore, CD20+ directed treatment of myeloma would complement chemotherapy by targeting chemoresistant clonogenic myeloma cells.

Previous studies showed that therapy with Rituximab, unlabeled anti-CD20 antibody, could be active in multiple myeloma (Hussein et al. 1999, Treon et al, 2002).

In this study, we propose to apply therapy with Bexxar, a radiolabeled anti-CD20 antibody. Bexxar Therapeutic Regimen is composed of the murine anti-CD20 monoclonal antibody Tositumomab and Iodine I 131 Tositumomab. Iodine I 131 Tositumomab is a radio-iodinated derivative of Tositumomab that has been covalently linked to Iodine-131.

We hypothesized that radiolabeled anti-CD20 antibody will be more efficacious than unlabeled antibody (i.e. rituximab) in eradication of highly radiosensitive myeloma cells, similarly to what was observed in non-Hodgkin's lymphoma (Horning et al., 2000; Davis et al, 2001 Flinn et al, 2001; Witzig et al, 2002). It is presumed, that higher efficacy of radiolabeled anti-CD20 antibody, if compared to unlabeled antibody, may be due to "crossfire effect" as the radiation is delivered not only to target cells but also to neighboring cells, both expressing and not-expressing CD20 (Vose et al, 1999). In the proposed design, we will apply Bexxar after completion of a course of initial chemotherapy for newly diagnosed patients or a course of salvage chemotherapy, provided that patients achieve at least partial response to prior therapy (i.e. > 50% reduction of tumor mass) and reach a plateau of their response to prior therapy. By using patients in a period of stable disease, we will have a better chance to observe the effects of radioimmunotherapy against CD20+ cells, which represent a minority of all malignant cells. In addition, we will evaluate the impact of Bexxar therapy on clonogenic myeloma cells using clonogenic assays as described in Methods.

We anticipate that majority of newly diagnosed patients will be eligible and will subsequently proceed to autologous stem cell transplant as part of standard therapy of myeloma (NCCN Guidelines 2004) if, as hypothesized, bexxar treatment does have the potential to eliminate clonogenic myeloma stem cells; stem cells collected post-bexxar treatment should be depleted of re-populating myeloma cells. Therefore, this combination of chemotherapy and targeted therapy against clonogenic cells may have a potential of eliminating myeloma clones. Although stem cell collections and autologous stem cell transplants have been used without apparent difficulties in the past in patients treated with anti-CD20 radio-conjugates (Ratanatharatorn et al, 2001; Kaminski et al, 2001; Ansell et al, 2002), we plan to collect backup stem cells prior to treatment with Bexxar, to allow to proceed with the standard stem cell transplant in the unlikely cases of failure of collection of stem cells post-Bexxar. Anti-CD20 radioimmunotherapy was previously used in combination with chemotherapy without additional toxicity (Emmanoulides et al, 2001; Gregory et al, 2001, Press et al, 2003).

Radioimmunotherapy of B-Cell Malignancies:

Radiolabeled monoclonal antibodies are efficacious in treating B-cell malignancies for the following reasons: B-lymphocytes, lymphoma, and myeloma cells are inherently sensitive to radiotherapy (Parker et al, 1980); the local emission of ionizing radiation by radiolabeled antibodies may kill cells with or without the target antigen in close proximity to the bound antibody; and penetrating radiation may obviate the problem of limited access in bulky or poorly vascularized tumors.

Early investigations of therapeutic radiolabeled antibodies for B-cell lymphoma were performed with iodinated antibodies (Press et al, 1989; Kaminski et al, 1993; Wahl et al, 1994; Press et al, 1995). Currently, two treatment regimens have been approved for treatment of relapsed/refractory and transformed follicular lymphoma. The Bexxar Treatment Regimen includes murine anti-CD20 antibody Tositumomab iodinated with Iodine I 131. The Main anti-tumor effect comes from high energy beta particles emitted by I 131. In addition, I 131 is emitting also low energy gamma radiation, allowing for gamma camera measurements and calculation of individualized dose of radioactive tracer for a given patient during therapeutic phase (see below). In Zevalin, a murine anti-CD20 antibody ibritumomab is covalently linked to 90Yttrium (90Y), which is a pure beta emitter. Lack of gamma radiation from 90Y does not allow for dosimetric assessments and a fixed dose of Zevalin is used for all patients based on their weight. This can possibly result in either under- or overdosing of some patients.

In addition to treatment of follicular lymphoma, ongoing studies explore a possibility of treatment with either Bexxar or Zevalin of other B-cell malignancies. In particular, anti-CD20 radioimmunotherapy appears very promising as part of treatment of mantle cell lymphoma, large cell lymphoma, and Waldenstrom's macroglobulinemia.

Iodine I 131 Tositumomab

Background:

Tositumomab is a murine IgG2a lambda monoclonal antibody directed against the CD20 antigen, which is found on the surface of normal and malignant B lymphocytes. Tositumomab is produced in an antibiotic-free culture of mammalian cells and is composed of two murine gamma 2a heavy chains of 451 amino acids each and two lambda light chains of 220 amino acids each. The approximate molecular weight of Tositumomab is 150 kD. In vitro studies have demonstrated that upon binding to the CD20 antigen, Tositumomab is capable of inducing apoptosis. In addition, Tositumomab induces antibody-dependent cellular cytotoxicity (ADCC) and complement-dependent cellular cytotoxicity (CDC). Iodine I 131 Tositumomab is a radio-iodinated derivative of Tositumomab that has been covalently linked to Iodine-131. Unbound radio-Iodine and other reactants have been removed by chromatographic purification steps. This agent produces its cytotoxic effect through the antitumor effects of ionizing radiation, as well as the more direct antitumor effects of the antibody. The goal of treatment with Iodine I 131 Tositumomab is selective delivery of radiotherapy to radiosensitive malignant cells, thus minimizing toxicity to the normal organs.

Bexxar Clinical Experience:

The dosing regimen and maximally tolerated dose of Bexxar were established in a phase I/II single-center study conducted at the University of Michigan (Kaminski et al, 2000). The RIT-II-001 trial included 47 patients and was designed to validate the dosing methodology developed at Michigan (Vose et al, 2000). The RIT-II-002 trial randomized 78 patients to receive either the tositumomab and I 131-tositumomab regimen or the unlabeled tositumomab to determine the value added of the radionuclide component (Davis et al, 2001). Patients treated on the radiolabeled antibody arm showed a higher overall response rate (OR = 55% vs. 19%) and complete response rate (CR = 33% vs. 8%). The RIT-II-004 study enrolled 60 patients with chemotherapy-refractory disease (no response or response lasting less than 6 months to the last chemotherapy received) to assess the efficacy of the Bexxar therapeutic regimen in this patient population (Kaminski et al, 2001). The number of patients who achieved longer duration of response to Bexxar was about 5 times higher than the number of patients who had a longer duration to chemotherapy (p <0.001). In addition, patients treated with Bexxar achieved a higher overall response (OR) rate (47% vs. 12%) and complete response (CR) rate (20% vs. 2%) than patients treated with chemotherapy. In summary, all 4 initial studies, including the Phase I/II trial, showed high response rates and duration of responses in patients with relapsed or refractory low grade or follicular lymphoma, including transformed follicular lymphoma previously-treated with chemotherapy. Most remarkably, patients who achieved complete responses experienced often particularly long duration of responses lasting for years. In recognition of remarkable activity, the FDA approved an expanded indication for the Bexxar Therapeutic Regimen on January 3, 2005.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Expected survival ≥ 6 months
* Pre-study performance status of 0, 1, or 2 according to the World Health Organization (WHO)
* Newly diagnosed or relapsed/refractory myeloma with histologic confirmation of multiple myeloma by the Department of Pathology at University of Michigan Cancer Center (UMCC)
* Not more than 3 lines of therapy for myeloma for patients with relapsed disease
* Documented Stage II or III multiple myeloma (Durie and Salmon, 1975) prior to initiation of first line therapy
* At least 4 cycles of first line (for newly diagnosed patients) or salvage (for relapsed/refractory patients) prior therapy and in a plateau of at least partial response (Blade et al, 1999) for at least 2 determinations 6 weeks apart
* At least 21 days from day 1 of the last cycle and fully recovered from all toxicities associated with prior surgery, radiation treatments, chemotherapy, or immunotherapy
* Measurable M-proteins with greater than 1 g/dl serum monoclonal protein and/or greater than 0.5 g/24 hour urine light chain excretion
* Acceptable hematologic status within two weeks prior to patient registration, including:

  * Absolute neutrophil count ([segmented neutrophils + bands] x total white blood cell [WBC]) ≥ 1,500/mm3;
  * Platelet counts ≥ 150,000/mm3; these patients will receive total body dose of 75 cGy of Bexxar; or
  * Platelet counts from 100,000/mm3 to 149,000/mm3; these patients will receive a 65 cGy total body dose of Bexxar;
  * In patients previously treated with ASCT, total body dose will be 55 cGy in patients with platelet count > 150,000 and 45 cGy in patients with platelets 100,000-149,000.
* Female patients who are not pregnant or lactating
* Men and women of reproductive potential who are following accepted birth control methods (as determined by the treating physician)
* Patients previously on Phase II drugs if no long-term toxicity is expected, and the patient has been off the drug for three or more weeks with no significant post treatment toxicities observed
* Patients determined to have < 25% bone marrow involvement with myeloma within six weeks of registration (based on bilateral core biopsy).

Exclusion Criteria:

* Patients with impaired bone marrow reserve, as indicated by one or more of the following:

  * Platelet count < 100,000 cells/mm3;
  * Hypocellular bone marrow;
  * Marked reduction in bone marrow precursors of one or more cell lines (granulocytic, megakaryocytic, erythroid);
  * History of failed stem cell collection;
  * Myelodysplastic syndrome (MDS) or evidence of other than myeloma clonogenic abnormalities;
  * Prior radioimmunotherapy;
  * Prior anti-CD20 therapy;
  * Other than myeloma malignancy, except B-cell non-Hodgkin's lymphoma, basal and squamous cell carcinoma of the skin, and cervical and breast cancer in situ, unless patient is cancer free for > 3 years;
  * Central nervous system (CNS) involvement;
  * Patients with known HIV infection;
  * Patients with pleural effusion;
  * Patients with abnormal liver function: total bilirubin > 2.0 mg/dL;
  * Patients with abnormal renal function: serum creatinine > 2.0 mg/dL;
  * Patients who have received prior external beam radiation therapy to > 25% of active bone marrow (involved field or regional);
  * Patients who have received G-CSF or GM-CSF therapy within two weeks prior to treatment;
  * Serious nonmalignant disease or infection which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives;
  * Major surgery, other than diagnostic surgery, within four weeks;
  * Presence of anti-murine antibody (HAMA) reactivity. This result must be available prior to receiving treatment for those patients with prior exposure to murine antibodies or proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-08; Primary Completion 2013-08 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kaminski, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bexxar Therapeutic
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bexxar Therapeutic
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 56 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With an Objective Response
Description: The primary objective is to determine of the rate of objective response (percentage of patients with an objective response) defined as sustained reduction of monoclonal proteins by more than 25% versus pre-Bexxar level.
  An objective response may be:
  Minimal Response (MR) - 25-49% reduction on the level of the serum monoclonal protein for at least 2 determinations.
  Partial Response (PR) - 50-89% reduction in the level of the serum monoclonal protein for at least 2 determinations.
  Complete Response (CR) - Absence of the original monoclonal protein in serum and urine on at least 2 determinations by immunofixation.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bexxar Therapeutic
Number analyzed (Participants) | 16
percentage of patients | 31 [11 to 59]

2. Secondary Outcome: Number of Participants With Complete Response (CR)
Description: Determine the rate of conversion to complete response (CR). CR requires all of the following:
  * Absence of the original monoclonal protein in serum and urine on at least 2 determinations by immunofixation. The presence of oligoclonal bands consistent with oligoclonal immune reconstitution does not exclude CR.
  * Less than 5% plasma cells in the bone marrow on at least 2 determinations. Repeat bone marrow is not required for patients with secretory myeloma who have sustained absence of monoclonal protein on immunofixation.
  * No increase in size or number of lytic bone lesions (development of a compression fracture does not exclude response).
  * Disappearance of all soft tissue plasmacytomas.
  * Patients in whom some, but not all the criteria for CR are fulfilled are classified as nCR or PR or VGPR (see below), providing the remaining criteria for nCR, VGPR, or PR are satisfied.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Bexxar Therapeutic
Number analyzed (Participants) | 16
participants | 2

3. Secondary Outcome: Duration of Response
Description: Progressive Disease (PD)-Free Interval (Duration of Response): measured, in a responder, from the date when a Complete Response, Complete Response, unconfirmed (CRu), or Partial Response (PR) is first noted to the first date at which progressive disease is observed. An ongoing PD-free interval occurs when there is a responder for whom progressive disease has not been noted.
Time Frame: up to approximately 15 years after treatment
Reporting Status: Not Posted

4. Secondary Outcome: Progression Free Survival Time
Description: Disease progression or death from Multiple Myeloma from start of study treatment
Time Frame: up to approximately 15 years after treatment
Reporting Status: Not Posted

5. Secondary Outcome: Time to Treatment Failure
Description: Of patients who initially responded (completely or partially) to treatment, at what subsequent point (measured in months) did they have progression of disease or begin a different treatment
Time Frame: up to approximately 15 years after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bexxar Therapeutic
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexxar Therapeutic (N=16)
Infection with Normal Neutrophil Count (Infections and infestations) | 1 (1)
Infection wtih Unknown Neutrophil Count (Infections and infestations) | 1 (1)
Neuropathy - Motor (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexxar Therapeutic (N=16)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 7 (7)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8 (10)
Platelets (Blood and lymphatic system disorders) | 9 (12)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2)
Pain - Other (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes